CLINICAL TRIAL: NCT03877757
Title: Evaluation of the Family Planning Elevated Statewide Contraceptive Service Delivery Initiative
Brief Title: Family Planning Elevated: Initiative Evaluation
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 117213
Record Dates: First submitted 2019-03-07; First posted 2019-03-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Contraception
Keywords: Family Planning; Implementation science; Evaluation; Contraceptive initiative

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family Planning Elevated Contraceptive Access Clinics Program: This group consists of community clinics who apply and are accepted for FPE CAP membership during the Family Planning Elevated initiative. These clinics will receive the intervention and will provide monthly service delivery data to the FPE evaluation team.
- Control Clinics: This group consists of non-participating community clinics matched on clinic size, geography, and client populations who are not interested in participating in the initiative but are willing to provide monthly service delivery data to the FPE evaluation team.

SUMMARY:
Family Planning Elevated (FPE) is a statewide contraceptive initiative with two primary aims: 1) supporting existing and proposed legislative policy that expands family planning services in Utah among low-income individuals covered by contraceptive legislation (currently individuals at ≤100% federal poverty) and 2) demonstrating additional existing service need among low-income individuals who currently fall in the contraceptive coverage gap (101%-250% federal poverty). Family Planning Elevated provides contraceptive grants, education and training, and technical assistance on comprehensive contraceptive care to participating clinics. The purpose of this evaluation is to assess the effect of FPE on clinic-level family planning service delivery among low-income women who fall in the contraceptive coverage gap compared to those receiving services from matched control clinics which did not receive the intervention. To assess these effects, FPE will collect monthly family planning service delivery data from both intervention and control clinics, beginning 12 months prior to the FPE intervention, and following for 12 months after the FPE intervention ends. A difference-in-difference analysis will compare trends and level-changes in family planning services provided to intervention and control groups.

DETAILED DESCRIPTION:
Intervention clinics (FPE Contraceptive Access Program [FPE CAP]) receive a multifaceted contraceptive intervention, including:

1. Training and technical assistance on contraceptive counseling and provision for FPE CAP providers, administrators, and health center support staff. FPE CAP staff will be required to attend an annual contraceptive training conference and receive additional remote and on-site technical support on counseling and provision of contraceptive methods. Methods include emergency contraception, oral contraceptive pills, contraceptive patch, vaginal ring, contraceptive injection, fertility awareness methods, condoms, contraceptive implant, hormonal IUDs, and non-hormonal IUD and other contraceptive methods, as feasible.
2. FPE will provide FPE CAP members a cash grant to offset personnel and equipment costs associated with FPE CAP start-up and implementation.
3. Monthly reimbursement for FPE CAP contraceptive services. As a result of the Medicaid Family Planning Waiver effective January 1, 2019, Utah health centers may claim Medicaid reimbursement for contraceptive services provided to Medicaid enrolled clients at ≤100% Federal Poverty Level. FPE CAP seeks to expand this coverage by providing reimbursement to FPE CAP health centers for contraceptive services provided to clients at 101% - 250% FPL (or 0% - 250% FPL for undocumented clients). Clients must be of reproductive age seeking female-user dependent methods and not be eligible for Medicaid/PCN.
4. Contraceptive method stock. The high upfront cost of some contraceptive methods, particularly IUDs and implants, is often a barrier for health centers to maintain adequate contraceptive inventory. During the FPE CAP project period, members will be provided a stock of IUDs and implants to provide to eligible FPE CAP clients. Health centers will be also be reimbursed or provided vouchers for short-acting methods including oral contraceptive pills, vaginal rings, contraceptive injections, condoms, cycle beads, and emergency contraception. FPE will provide technical assistance to members to build a sustainable inventory of contraceptive methods for the post-FPE CAP project period. This will include training on drug forecasting and stocking, 340B Drug Discount Program, group purchasing organizations, and patient assistance programs.
5. Evaluative Support: FPE CAP members will be responsible for providing routine data to FPE to help us assess the impact of the program. As part of this effort, FPE CAP members will receive evaluative support in developing and reporting data requirements both for the program and to fill existing clinical data needs around contraception. Additionally, data provided to the FPE team will be analyzed and returned back to the individual health centers as part of the dissemination strategy.
6. Marketing campaign: FPE will produce a targeted media campaign to increase public awareness of expanded eligibility for contraceptive services, improve demand for contraceptive services at community health centers, and provide client education on available contraceptive options. FPE will support FPE CAP members by creating customized media campaigns for community outreach and education.

Control clinics are similar clinics (matched by clinic size, geography, and serving Medicaid clients) who are not interested in participating in Family Planning Elevated, but are willing to provide the monthly service delivery data for the same time periods as their matched intervention clinic.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (age 18-50) who visited the intervention or control clinic within the allotted time frame.

Exclusion Criteria:

* Under age 18

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women of reproductive age
Study Population: The intervention occurs at the clinic level. Participating clinics are Utah health systems and individual clinics across Utah.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Change in total family planning services provided to women ages 18-49, as measured by monthly service delivery report | 12 months prior to FPE intervention start, for the 24-month intervention period, and for 12 months post-intervention
  Family planning services are defined as all family planning-related E/M, CPT, and HCPC codes within the FPE monthly service delivery report

SECONDARY OUTCOMES:
Changes in total long-acting reversible contraceptive services (LARC) provided to all women ages 18-49, as measured by monthly service delivery report | 12 months prior to FPE intervention start, for the 24-month intervention period, and for 12 months post-intervention
  Defined as all related E/M, CPT, and HCPC codes related to LARC methods within the FPE monthly service delivery report

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Simmons, PhD, Principal Investigator — University of Utah, Department of OBGYN
Locations (1):
- University of Utah, Department of Obstetrics & Gynecology, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen SR, Baayd J, Garcia G, Quade C, Gero A, Ekey M, Poggio C, Simmons R. Facility-based simulation as a programmatic tool for implementing a statewide contraceptive initiative. BMC Health Serv Res. 2022 Jul 29;22(1):965. doi: 10.1186/s12913-022-08332-4. PMID 35906656
- [Derived] Baayd J, Simmons RG. Protocol for a process evaluation of Family Planning Elevated: a statewide initiative to improve contraceptive access in Utah (USA). BMJ Open. 2020 Oct 1;10(10):e038049. doi: 10.1136/bmjopen-2020-038049. PMID 33004395